CLINICAL TRIAL: NCT03023319
Title: Phase I Study of the Non-receptor Kinase Inhibitor Bosutinib in Combination With Pemetrexed in Patients With Selected Metastatic Solid Tumors
Brief Title: Bosutinib in Combination With Pemetrexed in Patients With Selected Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nagla Abdel Karim (Other)
Responsible Party: Sponsor-Investigator, Nagla Abdel Karim, Associate Professor of Medicine, Augusta University
Organization: Augusta University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXP-16-01
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Mesothelioma; Bladder Cancer; Ovarian Cancer; Peritoneal Cancer; Thymoma; Thymus Cancer; Uterine Cervical Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma; Urinary Bladder Neoplasms; Ovarian Neoplasms; Thymoma; Thymus Neoplasms; Uterine Cervical Neoplasms | interventions — bosutinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Bosutinib and Pemetrexed (Experimental): Bosutinib and pemetrexed
  Interventions: Drug: Bosutinib; Drug: Pemetrexed

INTERVENTIONS:
Drug: Bosutinib — 100mg daily for 4 cycles (21 days per cycle)
Drug: Pemetrexed — 500 mg/m2 every 21 days for 4 cycles

SUMMARY:
This study will determine the maximum-tolerated dose (MTD) for oral bosutinib when used in combination with pemetrexed. The MTD is the highest dose of bosutinib with pemetrexed that can be given without causing severe side effects. This study will also test the safety of this combination and see what effects (good or bad) it has on participants and their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically proven advanced, metastatic non-squamous non-small cell lung cancer, pleural malignant mesothelioma, bladder or urethral cancer, ovarian cancer, primary peritoneal cancer, thymoma and thymic cancer and uterine cervical cancer.
* Measurable disease
* Life expectancy of greater than 3 months.
* Ability to take folic acid, vitamin B12, and dexamethasone according to protocol.

Exclusion Criteria:

- Untreated or symptomatic brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity of the combination of bosutinib and pemetrexed | 21 days
  CTCAE Grade 3 or 4 non-hematologic toxicities other than alopecia, nausea and vomiting.
Maximum tolerated dose of the combination of bosutinib and pemetrexed | completion of dose escalation

SECONDARY OUTCOMES:
Adverse events of the combination of bosutinib and pemetrexed | 16 weeks
Anti-tumor response rate | 6 and 12 weeks
Progression-free survival | 6 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nagla Karim, MD, Principal Investigator — Augusta University Georgia Cancer Center
Locations (1):
- Augusta University Georgia Cancer Center, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No